CLINICAL TRIAL: NCT05029817
Title: Ovarian Reserve in Women With Cystic Fibrosis and the Correlation With Demographic and Clinical Parameters
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Other Study IDs: HMO-0298-21
Record Dates: First submitted 2021-08-21; First posted 2021-09-01 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Cystic Fibrosis; Infertility, Female
Keywords: Antral follicular count; Anti-Mullerian hormone
MeSH Terms: conditions — Cystic Fibrosis; Infertility, Female

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main objective of this study is to assess the ovarian reserve of CF patients via measurement of AMH and AFC. Secondly, we aim to correlate between the ovarian reserve and demographic and clinical characteristics of these patients.

Outcomes measured will be levels of AMH and AFC, as compared to standard means in the general population. There is no need for a control group in this study since the standardized means of AMH and AFC in the general population are a more accurate comparable measure, which is based on data collected from large-scale populations, and thus accounts for confounding age factor in a more complete manner than can be obtained via a control group (Almog et al., 2011, La Marca et al., 2012, Penzias et al., 2020).

ELIGIBILITY:
Inclusion Criteria:

* Female patients diagnosed with CF according to genetic testing.
* Age 18-45 years old.
* Routinely attended the CF Center at Hadassah Medical Center.

Exclusion Criteria:

* Refusal to participate in the study.
* Age under 18 or above 45.
* Use of hormonal contraceptives (for the purpose of AFC).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Female CF patients seen regularly in the Hadassah Mt. Scopus CF Center, aged 18-45 years old, who regularly attended the clinic, and from whom demographic and clinical parameters are available.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-07-15 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
AMH levels | 24 hours
  Levels of Anti-Mullerian hormone
Antral follicular count | Through study completion, an average of 1 year.
  Antral follicular count as assessed by ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Anat Hershko Klement, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel, Jerusalem, Israel